CLINICAL TRIAL: NCT01912742
Title: Effect of Speed of Weight Loss on Compensatory Mechanisms Activated During Weight Reduction
Acronym: FVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Monash University (Other); Portuguese Research Council (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/888
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Obesity
Keywords: Weight loss; Speed of weight loss; Metabolic compensation; Diet therapy
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid weight loss group (Experimental): The rapid weight loss group will follow a commercial very-low calorie diet (VLCD) during 4 weeks. The participants allocated to this group will follow a 550 (women) - 660 (men) kcal/day diet. The VLCD products provide 110kcal/pack and include a variety of milkshakes, smoothies and soups. In addition to VLCD products, calorie-free drinks and some low-starch vegetables (maximum 2 cups/day) will be allowed. Drinking at least 2.5 liters of non-caloric liquids will be recommended.
  Interventions: Behavioral: Very-low calorie diet (VLCD)
- Slow weight loss group (Experimental): The slow weight loss group will be prescribed an individualized low calorie diet (LCD) (1200-1500kcal/day), during 8 weeks, using meal replacements (such as smoothies, soups and cereal bars) and conventional foods. The macronutrient composition will be matched with that of the VLCD.
  Interventions: Behavioral: Low calorie diet (LCD)

INTERVENTIONS:
Behavioral: Very-low calorie diet (VLCD)
  Arms: Rapid weight loss group
Behavioral: Low calorie diet (LCD)
  Arms: Slow weight loss group

SUMMARY:
Obesity has become a global epidemic with huge public health implications. Although clinical significant weight loss (WL) can be achieved by a combination of diet and behavioral modification, strong metabolic adaptations, with increased appetite and suppressed energy expenditure, are activated, which compromise WL maintenance and increase the risk of relapse. The aim of this project is to investigate the potential role of WL rate in modulating such responses. More specifically, the investigators want to determine if a similar WL achieved rapidly vs slowly induce the same compensatory responses to weight reduction. A secondary aim is to assess if speed of weight loss can influence motivation. A large battery of assessments will be performed before and after weight reduction including body composition, resting metabolic rate, substrate oxidation, exercise efficiency, fasting and postprandial release of several appetite-regulating hormones, subjective feelings of hunger and fullness and motivation. This project can bring large practical benefits concerning the design of weight loss programs to minimize weight relapse.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-50 years old)
* Obese healthy volunteers (30<BMI<45 kg/m2)
* Weight stable on the last three months (<2kg), not currently dieting to lose weight and with an inactive lifestyle)

Exclusion Criteria:

* History of endocrine/cardiovascular/pulmonary/kidney disease, anaemia, gout, milk intolerance, depression or other psychological disorders, eating disorders, drug or alcohol abuse within the last two years and current medication known to affect appetite or induce weight loss. Those with a planned surgery during the study period or participating in another research study will also not be accepted to take part in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Appetite related hormones | Before the start of the study and again at week 2 and 4 (VLCD group) and 4 and 8 (LCD group). And also, on week 12 (for both groups).
  Appetite-related hormones (active ghrelin, PYY, GLP-1, CCK) will be measured in fasting and every 30 minutes up to 2,5 hours
Body composition | Baseline, 2 and 4 weeks (VLCD group) and 4 and 8 weeks (LCD group) and 12 weeks (both groups)
  Body composition measured by air displacement plethysmography

SECONDARY OUTCOMES:
Resting metabolic rate (RMR) | Baseline, 2 and 4 weeks (VLCD group) and 4 and 8 weeks (LCD group) and 12 weeks (both groups)
  RMR measured by indirect calorimetry
Exercise efficiency | Baseline, 2 and 4 weeks (VLCD group) and 4 and 8 weeks (LCD group) and 12 weeks (both groups)
  Exercise efficiency measured by graded exercise on a bike

CONTACTS AND LOCATIONS:
Overall Officials: Bård Kulseng, MD PhD, Study Director — Norwegian University of Science and Technology; Catia Martins, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Coutinho SR, With E, Rehfeld JF, Kulseng B, Truby H, Martins C. The impact of rate of weight loss on body composition and compensatory mechanisms during weight reduction: A randomized control trial. Clin Nutr. 2018 Aug;37(4):1154-1162. doi: 10.1016/j.clnu.2017.04.008. Epub 2017 Apr 25. PMID 28479016